CLINICAL TRIAL: NCT00986895
Title: A Study of Glyceryl Tri-(4-phenylbutyrate) Administered Orally as a Single Dose, and Twice Daily for Seven Consecutive Days to Subjects With Hepatic Impairment With Cirrhosis and to a Control Group
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Collaborators: Ucyclyd Pharma, Inc. (Other)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: UP 1204-002
Record Dates: First submitted 2009-09-15; First posted 2009-09-30 (Estimated); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Hepatic Encephalopathy; Urea Cycle Disorders
Keywords: HPN-100; GT4P; Glyceryl tri-(4-phenylbutyrate)
MeSH Terms: conditions — Hepatic Encephalopathy; Urea Cycle Disorders, Inborn | interventions — glycerol phenylbutyrate

INTERVENTIONS:
Drug: HPN-100 — HPN-100 is a triglyceride that has a similar mechanism of action as NaPBA. It is a liquid with minimal taste and odor. HPN-100 is broken down to phenylbuteric acid (PBA). PBA is converted to phenylacetic acid (PAA) that is the active metabolite. Three teaspoons of HPN-100 (~17.4mL) delivers an equivalent amount of PBA to40 tablets of NaPBA.

SUMMARY:
The purpose of this study is to determine the safety and tolerability of GT4P administered orally as a single dose, and twice daily for 7 consecutive days, to subjects with hepatic impairment with cirrhosis (Child-Pugh scores of A, B, or C) and to a gender matched and similar age control group with normal hepatic function.

DETAILED DESCRIPTION:
Study acquired from Horizon in 2024.

ELIGIBILITY:
Inclusion Criteria:

Subjects were required to fulfill the following criteria in order to participate in the study:

Screening:

* Males or females aged ≥ 18 years of age
* Able to provide written informed consent before any study-related procedures, and ability, in the opinion of the Investigator, to comply with all the requirements of the study
* Classification to one of the following:

  * current diagnosis of hepatic impairment with cirrhosis
  * healthy subject
* Subjects with hepatic impairment with cirrhosis were classifiable to one of the following groups:

  * Child-Pugh score A
  * Child-Pugh score B
  * Child-Pugh score C
* Subjects with hepatic impairment with cirrhosis who were on a therapeutic regimen of lactulose must have been on a stable dose for ≥ 30 days prior to screening
* If female, a negative pregnancy test at screening and pre-dose on day 0, or a documented sterilization procedure; a female of child-bearing potential must have been using a medically approved birth control method and must have agreed to use the same method of contraception during the full course of the study (on pre-dose day 0 as well as at screening)
* Weight within the range of 60-100 kg (at screening and pre-dose on day 0)
* Willing to stop taking any medication that the Sponsor and the Investigator felt was not appropriate for use during the study, beginning 2 days before dosing and throughout the study

Exclusion Criteria:

Subjects who fulfilled any of the following criteria were excluded from the study:

Screening:

* Clinically significant history or evidence of cardiovascular, respiratory, renal, gastrointestinal, endocrine, neurological, immunological, or psychiatric disorder(s), as determined by the Investigator
* Serum sodium < 120 mEq/L
* Serum creatinine ≥ 1.5 upper limit of normal
* Potassium ≤ 3.5 mEq/L
* Other laboratory values outside the normal range which were determined to be clinically significant by the Investigator
* Significant illness within the last 14 days
* Oral temperature > 38.5°C or < 36°C and/or a suspected site of active infection
* Inflammatory bowel disease or malabsorption defined with steatorrhea
* Active gastrointestinal bleeding, defined as melena, hematochezia, or hematemesis requiring hospitalization within the last 30 days
* Use of probenecid, valproate, or corticosteroids within the last 24 hours
* Use of any medication, other than those approved by the Sponsor and Investigator, in the last 48 hours
* History of seizures within the last 72 hours
* Positive drugs of abuse urine test
* Positive alcohol breath test
* Donation or loss of blood (500 mL or more) within the last 30 days
* Donation or loss of plasma within the last 7 days
* History of acquired immunodeficiency syndrome (AIDS) or determined human immunodeficiency virus (HIV) positive
* Hepatitis B or C (HBV; HCV) positive (healthy volunteers only)
* Use of any investigational drug within the last 30 days
* Known hypersensitivity to sodium phenylbutyrate or similar drugs
* Emergency hospitalization within the last 90 days
* Intake of alcohol in the last 7 days

Pre-dose (days 0 and 7):

* Significant illness or emergency hospitalization since the last study visit
* Oral temperature > 38.5°C or < 36°C and/or a suspected site of active infection
* Use of probenecid, valproate, or corticosteroids within the last 24 hours
* Use of any non-approved medication (by the Sponsor/Investigator) within the 48 hours before dosing
* History of seizures within the last 72 hours
* Positive drugs of abuse urine test
* Positive alcohol breath test
* Donation or loss of blood (500 mL or more) or plasma since the last study visit
* Use of any investigational drug since the last study visit
* Intake of alcohol in the last 7 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2006-09; Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
The rate of adverse event

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (2):
- Ukraine (2):
  - National University of Pharmacy, Kharkiv
  - Department of General Surgery #2; Kharkiv State Medical University, Kharkiv

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- [Derived] McGuire BM, Zupanets IA, Lowe ME, Xiao X, Syplyviy VA, Monteleone J, Gargosky S, Dickinson K, Martinez A, Mokhtarani M, Scharschmidt BF. Pharmacology and safety of glycerol phenylbutyrate in healthy adults and adults with cirrhosis. Hepatology. 2010 Jun;51(6):2077-85. doi: 10.1002/hep.23589. PMID 20512995